CLINICAL TRIAL: NCT04297956
Title: Survey on Patients After Childbearth Following Bariatric Surgery - Data Collection on Mental Health Complications, Weight Change, Nutrition Deficiencies and Postpartal Progress
Brief Title: Survey on Patients After Childbearth Following Bariatric Surgery
Acronym: SPOtMom
Status: Completed | Type: Observational
Sponsor: Wuerzburg University Hospital (Other)
Responsible Party: Principal Investigator, Ann-Cathrin Koschker, Head of outpatient clinic for diabetes and lipids, Wuerzburg University Hospital
Other Study IDs: spot_mom
Record Dates: First submitted 2020-02-24; First posted 2020-03-06 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Bariatric Surgery Status in Childbirth; Puerperal Depression
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Women with a history of bariatric surgery may face various difficulties during pregnancy and puerperal time. Therefore it is assumed the prevalence of mental health disorders might be higher than in average women during and after pregnancy. This could possibly lead to an unsatisfying weight progress and therapeutic non-adherence. These factors shall be observed in the study in order to characterize this special cohort of participants.

DETAILED DESCRIPTION:
Women following bariatric surgery are included at least 6 months after childbirth to evaluate retrospectively pregnancy and puerperal time. For mental health issues questionnaires, a structured clinical interview (SCID) and a psychological interview give an insight to past and present status. In order to evaluate weight progress and nutrient deficiencies routine follow-up care data of bariatric surgery is screened. In order to assess the course of pregnancy and child development data is extracted from pregnancy and child's examinations reports. Furthermore medication adherence, quality of life and sleep are registered by questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* status following bariatric / metabolic surgery due to indication criteria
* childbirth after bariatric / metabolic surgery, at least 6 months ago
* written informed consent

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Patients visiting the metabolic ambulance for follow-up care after bariatric surgery are eligible for the study.
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Number of patients with prevalence of symptoms of depression or anxiety assessed by questionnaires and structured clinical interview (SCID) | date of recruitement (> 6 months after childbirth)
  questionnaires for depression:
  * Beck Depression Inventory (BDI-II)
  * Patient Health Questionnaire-9 (PHQ-9)
  * Edinburgh Postnatal Depression Scale (EPDS)
  questionnaire for anxiety:
  * Generalized Anxiety Disorder-7 (GAD-7)
  Prevalence of symptoms can be defined by scores higher than defined cut-offs in questionnaires or scores that lead to diagnosis of psychiatric disorder in structured clinical interview
Number of patients with prevalence of symptoms of depression or anxiety assessed by questionnaires and structured clinical interview | retrospective: time frame 0-4 weeks after birth
  questionnaires for depression:
  * Patient Health Questionnaire-9 (PHQ-9)
  questionnaire for anxiety:
  * Generalized Anxiety Disorder-7 (GAD-7)
  Prevalence of symptoms can be defined by scores higher than defined cut-offs in questionnaires or scores that lead to diagnosis of psychiatric disorder in structured clinical interview
Number of patients with prevalence of symptoms of depression assessed by structured clinical interview | retrospective: complete lifetime from date of birth until date of recruitment (> 6 months after childbirth), assessed up to 50 years
  Prevalence of symptoms can be defined by scores that lead to diagnosis of psychiatric disorder in structured clinical interview

SECONDARY OUTCOMES:
Mean change of body weight from baseline | from date of bariatric surgery until date of recruitment (> 6 months after childbirth), assessed up to 20 years
  Body weight is measured on scales and participants are asked additionally via questionnaire. Baseline measurement starts at date of bariatric surgery.
Status of nutritional deficiencies and therapy adherence | from date of bariatric surgery until date of recruitment (> 6 months after childbirth), assessed up to 20 years
  Participants are asked to answer Medication Adherence Report Scale (MARS-D) and blood levels concerning nutrients that are examined routinely in bariatric surgery follow-up care are analysed.
Adverse events in pregnancy and child development | from date of beginning of pregnancy until date of recruitment (> 6 months after childbirth), assessed up to 12 years
  Record of prenatal care and record of child's examinations are screened for complications.

CONTACTS AND LOCATIONS:
Overall Officials: Ann-Cathrin Koschker, Dr. med., Principal Investigator — Würzburg University Hospital
Locations (5):
- Germany (5):
  - University Hospital, Würzburg, Bavaria
  - Sana Adipositaszentrum Offenbach, Offenbach, Hesse
  - Uniklinikum Aachen, Klinik für Allgemein-, Viszeral-und Transplantationschirurgie, Aachen, North Rhine-Westphalia
  - Sana Adipositaszentrum NRW, Remscheid, North Rhine-Westphalia
  - Adipositaszentrum Westküstenklinium Heide, Heide, Schleswig-Holstein